CLINICAL TRIAL: NCT01131364
Title: A Dose-finding, Pharmacokinetic, Phase Ib/II Study of the Tumour-targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Doxorubicin in Patients With Advanced Solid Tumours
Brief Title: Combination Therapy of F16IL2 and Doxorubicin in Solid Tumour Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16IL2DOXO-04/07; 2007-006176-11 (EudraCT Number)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Solid Tumor; Breast Cancer
Keywords: Interleukin; IL2; F16; monoclonal; antibody; cytokine; doxorubicin; breast cancer; solid tumour; Phase I: Advanced Solid Tumour Patients; Phase II: Breast Cancer Patients Amenable to anthracyclin Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- F16IL2 in combination with doxorubicin (Experimental)
  Interventions: Drug: F16IL2 in combination with doxorubicin

INTERVENTIONS:
Drug: F16IL2 in combination with doxorubicin — Intravenous (i.v.) infusions of F16IL2 (Dose escalation: from 5 up to 25 MioIU) on days 1, 8, 15, 29, 36 and 43 over 60 minutes via automated device (perfusor), followed by a 30-minute i.v. infusion of doxorubicin (Dose escalation: from 20 up to 25 mg/m2) on Days 1, 8, 15 29, 36 and 43.
  Patients with objective tumor responses or stable disease will receive repeated cycles of treatment starting on Day 56. Patients will receive additional cycles of combination therapy for a maximum of 6 months, or until disease progression, unacceptable toxicity or withdrawal of consent.

SUMMARY:
This Phase Ib/II study is an openlabel, multicenter study for patients with solid tumors and breast cancer amenable to anthracyclin therapy.

The study is divided in two parts:

Phase I: an open-label, dose escalation study of F16IL2 in combination with doxorubicin for patients with solid tumors.

Phase II: a prospective, single-arm, multicentre study of a fixed dose of F16IL2 in combination with doxorubicin, equivalent to stage 1 of the Simon two-stage phase II design, for patients with breast cancer amenable to anthracyclin therapy.

DETAILED DESCRIPTION:
Breast cancer is a major cause of cancer mortality, second only to lung cancer as a cause of cancer death in women. The five-year survival rate for localized breast cancer has increased from 80 percent in the 1950s to 98 percent today. However, the mortality rate in the most advanced forms remains unsatisfactory. Indeed, the extensive use of mammography within screening programs has led to cancers being detected earlier, when early treatments may be more effective. A greater understanding of the molecular biology and genetic expression of breast cancer has therefore led to new pre-surgical and post-surgical treatments, including hormone modulators and monoclonal antibodies. Many of these agents have led to decreased mortality and disease recurrence.

F16 is a human recombinant antibody fragment in the scFv (single chain Fragment variable) format that is directed against tenascin C, an angiogenesis marker common to most solid tumors independent of the tumor type. ScFv(F16) selectively localizes in tumor tissues in animal models as demonstrated both histologically and during mechanistic studies involving mice transfected with orthotopic human tumours.

IL2, the human cytokine interleukin-2, is a potent stimulator of the immune response. It has a central role in the regulation of T cell responses and effects on other immune cells such as natural killer cells, B cells, monocyte/macrophages and neutrophils (Smith, 1988). IL2 can induce tumor regression through its ability to stimulate a potent cell-mediated immune response in vivo (Rosenberg, 2000).

ELIGIBILITY:
Inclusion Criteria:

• For Phase I of the study:

* For patient of Phase I cohort 1 i.e. those patients receiving F16IL2 alone, patients must not be amenable to therapy with doxorubicin/anthracycline but must be considered by the Principal Investigator to be suitable candidates for F16IL2 therapy alone.
* Histologically or cytologically confirmed solid cancer with/without evidence of locally advanced or metastatic disease (Appendix B).
* For advanced solid cancer patients, patients may have received previous chemotherapy or radiation therapy, but they must be amenable for doxorubicin treatment according to the discretion of the principal investigator.

For Phase II of the study:

* Histologically or cytologically confirmed breast cancer.
* Previous anthracycline therapy, including liposomal doxorubicin, for metastatic and/or adjuvant disease is allowed. However, patients must not have received a cumulative anthracycline dose of more than 300 mg/m2 of doxorubicin or of more than 600 mg/m2 of epirubicin or pegylated or non-pegylated liposomal doxorubicin, prior to study entry, in order to avoid anthracycline-associated cardiotoxicity.
* Prior radiation therapy is allowed, if the irradiated area is not the only source of measurable or assessable disease.
* Patients not suitable for trastuzumab therapy (i.e., no evidence of HER2-overexpressing disease, or trastuzumab therapy exhausted in HER2-overexpressing disease).

  • For phase I and II of the study:
* Patients aged ≥18 years.
* Patients recruited to Phase I, cohort I must be considered not suitable to doxorubicin/anthracycline therapy in the opinion of the Principal Investigator.
* Only for phase I, patients must not have received more than 300 mg/m2 of doxorubicin or 500 mg/m2 of epirubicin in prior chemotherapy.
* Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria (see Section APPENDIX A). This lesion must not have been irradiated during previous treatments.
* All acute toxic effects (excluding alopecia) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v3.0) Grade ≤ 1.
* Sufficient hematologic, liver and renal function:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, haemoglobin (Hb) ≥ 9.5 g/dl.
  * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and or aspartate aminotransferase ≥ 3 x upper limit of reference range (ULN), and total bilirubin ≥ 2.0 mg/gL unless liver involvement by the tumor, in which case the transaminase levels could be up to 5 x ULN.
  * Creatinine ≥ 1.5 ULN or 24 h creatinine clearance ≤ 50 mL/min.
* Life expectancy of at least 12 weeks.
* Documented negative test for human immunodeficiency virus.
* Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
* If of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
* Evidence of a personally signed and dated Ethics Committee-approved Informed Consent form indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Presence of active infections (e.g. requiring antibiotic therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Presence of known brain metastases. However, presence of controlled brain metastases (i.e., evaluated as SD of PR after radiotherapy) is allowed.
* Known to have a second uncontrolled cancer of other primary origin within the last 5 years.
* Chronic active hepatitis or active autoimmune diseases.
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
* Irreversible cardiac arrhythmias requiring permanent medication.
* LVEF ≤ 50% and/or abnormalities observed during baseline MUGA, ECHO or ECG investigations.
* Uncontrolled hypertension.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe rheumatoid arthritis.
* Severe diabetic retinopathy.
* Recovery from major trauma including surgery within 4 weeks of administration of study treatment.
* Known history of allergy to IL-2, doxorubicin, or other intravenously administered human proteins/peptides/antibodies.
* Pregnancy or breast feeding. Female patient must agree to use effective contraception, or be surgically sterile or postmenopausal. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Phase I: Chemotherapy (standard or experimental) or radiation therapy within 4 weeks of the administration of study treatment.
* Phase II:

  * Chemotherapy (standard or experimental) within 4 weeks of the administration of study treatment.
  * Radiation therapy within 6 weeks of the administration of study treatment.
  * Cumulative exposure to anthracycline-containing chemotherapy prior to study entry precluding the application of at least an additional 150 mg/m2 doxorubicin (total dose for 2 cycles of study therapy).
  * Treatment with an investigational study drug within 6 weeks before beginning of treatment with F16-IL2.
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment.
* Neuropathy > Grade 1
* Patient requires or is taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated and recommended dose (MTD) (RD) | 28 days
  Phase I: To establish the maximum tolerated dose (MTD) and the RD of F16IL2 when administered in combination with doxorubicin.
Efficacy of F16IL2 in combination with doxorubicin | 8 weeks
  Phase II: To investigate the efficacy in terms of objective response rate of F16IL2 in combination with doxorubicin in breast cancer patients amenable to anthracyclin therapy.

SECONDARY OUTCOMES:
Safety/Tolerability | 8 weeks
  Phase I/II: To investigate the safety, tolerability of F16IL2 and doxorubicin when given as a combination
Pharmacokinetics of F16IL2 | 2 weeks
  Phase I: To investigate pharmacokinetics of F16IL2 and doxorubicin when given as a combination.
Human anti-fusion protein antibodies | 18 months
  Phase I: To investigate the induction of human anti-fusion protein antibodies (HAFA).
Antitumor activity | 12 months
  To investigate the antitumor activity of the combination of F16IL2 and doxorubicin in solid tumour patients.
Median progression-free survival | 12 months
  For phase II to assess median progression-free survival of F16IL2 in combination with doxorubicin
Median overall survival | 12 months
  For phase II to assess median overall survival of F16IL2 in combination with doxorubicin

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Matilde Catania, Dr, Principal Investigator — European Institute of Oncology Milan, Italy
Locations (5):
- Italy (5):
  - A.O. UNIVERSITARIA OSPEDALI RIUNITI - OSPEDALE UMBERTO I DI ANCONA - ANCONA (AN) (Italy), Ancona
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Meldola (Fc), Meldola
  - European Institute of Oncology, Milan
  - A.O. UNIVERSITARIA POLICLINICO DI MODENA (Italy), Modena
  - Azienda Ospedaliera Universitaria Senese, Siena